CLINICAL TRIAL: NCT02147613
Title: High-intensity Aerobic Interval Training vs. Moderate-intensity Continuous Exercise Training in Heart Failure With Preserved Ejection Fraction
Brief Title: High Intensity Interval Exercise in Diastolic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Mayo Clinic (Other); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mayo-ArizonaSU Seed 93016001
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-01

CONDITIONS: Diastolic Heart Failure
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- High intensity interval training (Experimental): High intensity interval training - 3 days per week at 85-90% peak heart rate (4x4 bouts) for 1 month (12 sessions of exercise)
  Interventions: Other: High intensity interval training
- Moderate intensity exercise training (Active Comparator): 3 days/week, 30 mins at 70% Peak heart rate for 1 month (12 sessions of exercise)
  Interventions: Other: Moderate intensity exercise training

INTERVENTIONS:
Other: High intensity interval training — 3 days per week at 85-90% peak heart rate (4x4 bouts) for 1 month (12 sessions of exercise)
  Arms: High intensity interval training
Other: Moderate intensity exercise training — 3 days/week, 30 mins at 70% Peak heart rate for 1 month (12 sessions of exercise)
  Arms: Moderate intensity exercise training

SUMMARY:
Heart failure is a major health concern and is the leading cause of hospitalization among elderly Americans. Currently 5.7 million Americans are estimated to have heart failure and the estimated direct and indirect costs of treating heart failure are approximately $37.2 billion. Approximately 40% of those diagnosed with heart failure will have heart failure with preserved ejection fraction (HFPEF). These individuals have significant restrictions in their ability to carry out activities of daily living. Exercise training has been established as adjuvant therapy in heart failure. Although exercise training guidelines for treatment of heart failure with reduced ejection fraction (HFREF) are well established, no consensus exercise guidelines exist for management of HFPEF. Aerobic and cardiovascular adaptations are generally greater after high-intensity exercise training; interval-type exercise facilitates this type of training because it allows for rest periods that make it possible for patients with heart failure to perform short (e.g., 1-4 minutes) work periods at intensities that are higher than would be possible during continuous exercise. High-intensity aerobic interval training presents a unique, yet untested, therapeutic modality for the exercise training of patients with heart failure with preserved ejection fraction. Pilot testing is warranted, results of which may have important implications for reducing cardiovascular risk, increasing short- and long-term quality of life and survival, and reducing healthcare costs in this patient population. The investigators primary specific aim is to determine the efficacy of a novel, high-intensity aerobic interval exercise training program for improving VO2peak (peak oxygen uptake), endothelial function, and arterial stiffness in patients with HFPEF. The investigators secondary aim is to determine whether the vascular changes are correlated with the changes in VO2peak.

DETAILED DESCRIPTION:
Heart failure is a major health concern and is the leading cause of hospitalization among elderly Americans. Currently 5.7 million Americans are estimated to have heart failure and the estimated direct and indirect costs of treating heart failure are approximately $37.2 billion. Approximately 40% of those diagnosed with heart failure will have heart failure with preserved ejection fraction (HFPEF).2 These individuals have significant restrictions in their ability to carry out activities of daily living.

Exercise training has been established as adjuvant therapy in heart failure.4 Although exercise training guidelines for treatment of heart failure with reduced ejection fraction (HFREF) are well established, no consensus exercise guidelines exist for management of HFPEF. Exercise training increases VO2peak, thus improving prognosis for patients with heart failure. Indeed, VO2peak has been reported to be the single best predictor of mortality in those with cardiac disease.6 Exercise training also improves endothelial function and reduces arterial stiffness, as well as enhancing quality of life.7,8 Because HFPEF is associated with a both diastolic dysfunction and a loss of compensatory systemic vasodilator reserves, arterial stiffness and endothelial function are especially important in this population.

Aerobic and cardiovascular adaptations are generally greater after high-intensity exercise training; interval-type exercise facilitates this type of training because it allows for rest periods that make it possible for patients with heart failure to perform short (e.g., 1-4 minutes) work periods at intensities that are higher than would be possible during continuous exercise. For example, Wisloff et al. demonstrated the superiority of high-intensity aerobic interval training, as compared to continuous, moderate-intensity exercise training, in patients with stable postinfarction heart failure (with reduced ejection fraction). Not only was VO2peak and FMD improved more, patients tolerated the high-intensity program without reported incident. Furthermore, they found it "motivating to have a varied procedure to follow," whereas patients found the continuous exercise group training sessions to be "quite boring." High-intensity aerobic interval training presents a unique, yet untested, therapeutic modality for the exercise training of patients with heart failure with preserved ejection fraction.

Pilot testing is warranted, results of which may have important implications for reducing cardiovascular risk, increasing short- and long-term quality of life and survival, and reducing healthcare costs in this patient population.Patients undergoing exercise training live on average 2.16 years longer at the extremely low cost-effectiveness ratio of $1494 per life year saved.Since the majority of this patient population belongs to the Medicare age group, this intervention has significant potential to reduce healthcare costs.

Hypotheses and Specific Aims Our primary specific aim is to determine the efficacy of a novel, high-intensity aerobic interval exercise training program for improving VO2peak, endothelial function, and arterial stiffness in patients with HFPEF. Our secondary aim is to determine whether the vascular changes are correlated with the changes in VO2peak.

We hypothesize that improvements in VO2peak, endothelial function, and arterial stiffness will be greater after the high-intensity aerobic interval training program and that vascular adaptations will be correlated with changes in VO2peak.

ELIGIBILITY:
Inclusion Criteria:

* HFpEF diagnosis with New York Heart Association heart failure Class II-III symptoms

Exclusion Criteria:

* Unstable angina
* Myocardial infarction in the past 4 weeks
* Uncompensated heart failure
* New York Heart Association class IV symptoms
* Complex ventricular arrhythmias (at rest or during the maximal exercise test)
* Medical or orthopedic conditions that precluded treadmill walking
* Symptomatic severe aortic stenosis
* Acute pulmonary embolus
* Acute myocarditis
* Medication non-compliance

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arizona State University, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona

REFERENCES:
- [Derived] Angadi SS, Mookadam F, Lee CD, Tucker WJ, Haykowsky MJ, Gaesser GA. High-intensity interval training vs. moderate-intensity continuous exercise training in heart failure with preserved ejection fraction: a pilot study. J Appl Physiol (1985). 2015 Sep 15;119(6):753-8. doi: 10.1152/japplphysiol.00518.2014. Epub 2014 Sep 4. PMID 25190739

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Intensity Interval Training | Moderate Intensity Exercise Training
Started | 10 | 9
Completed | 9 | 6
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Intensity Interval Training | Moderate Intensity Exercise Training | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants] — Population: Subjects who completed
  Participants
    number analyzed (Participants) | 9 | 6 | 15
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 2 | 1 | 3
    >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Mean age of participants that completed the study
  years
    Mean age of completers: number analyzed (Participants) | 9 | 6 | 15
    Mean age of completers | 69 (6.1) | 71.5 (11.7) | 69.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Composition of participants that completed
  Participants
    number analyzed (Participants) | 9 | 6 | 15
    Female | 1 | 2 | 3
    Male | 8 | 4 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Diastolic Dysfunction
Description: Measured using left ventricular echocardiography. Diastolic dysfunction is graded as: normal, grade 1, grade 2, grade 3, grade 4. Increasing grade is indicative of worsening LV dysfunction and worse outcomes. Improvement in LV grade is associated with better long term outcomes.
Time Frame: Before and after the 1 month exercise intervention
Measure: Mean (Standard Deviation); unit: DD grade
Arm/Group | High Intensity Interval Training | Moderate Intensity Exercise Training
Number analyzed (Participants) | 9 | 6
DD grade
  Pre | 2.1 (0.3) | 2 (0.6)
  Post | 1.3 (0.7) | 2.2 (0.8)

2. Secondary Outcome: VO2peak
Description: Measured using a graded exercise test (modified Bruce protocol) with 12-lead EKG monitoring and ventilatory gas exchange analysis.
Time Frame: Test carried out before and after the 1 month long exercise intervention.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | High Intensity Interval Training | Moderate Intensity Exercise Training
Number analyzed (Participants) | 9 | 6
ml/kg/min
  Pre | 19.2 (5.2) | 16.9 (3)
  Post | 21 (5.2) | 16.8 (4)

3. Other Pre Specified Outcome: Brachial Artery Flow-mediated Dilation
Description: Reactive hyperemia mediated brachial artery dilation will be measured after 5 minutes of ischemia with forearm cuff occlusion. Artery will be continuously monitored using B-mode ultrasound.
Time Frame: Before and after 1-month exercise intervention
Measure: Mean (Standard Deviation); unit: percentage of FMD
Arm/Group | High Intensity Interval Training | Moderate Intensity Exercise Training
Number analyzed (Participants) | 9 | 6
percentage of FMD
  Pre | 6.9 (3.7) | 8.1 (4.1)
  Post | 7 (4.2) | 3.4 (3.6)

ADVERSE EVENTS:
Arm/Group | High Intensity Interval Training | Moderate Intensity Exercise Training
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes